CLINICAL TRIAL: NCT07078604
Title: A Phase II Trial of the Immunogenicity of a DNA Plasmid-Based Vaccine (STEMVAC) Encoding Th1 Selective Epitopes From Five Antigens Associated With Breast Cancer Stem Cells (MDM2, YB1, SOX2, CDH3, CD105) in Patients With Metastatic Triple-Negative Breast Cancer
Brief Title: A Cancer Vaccine (STEMVAC) in Combination With Chemotherapy for the Treatment of PD-L1 Negative Metastatic Triple-Negative Breast Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Kuni Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RG1125414; NCI-2025-04327 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 20925 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2025-07-11; First posted 2025-07-22 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-09

CONDITIONS: Anatomic Stage IV Breast Cancer AJCC v8; Metastatic Triple-Negative Breast Carcinoma
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — Cisplatin; 1,2-diaminocyclohexaneplatinum II citrate; Platinum; Docetaxel; Doxorubicin; eribulin; Paclitaxel; Taxes; liposomal doxorubicin; sargramostim; Colony-Stimulating Factors; Carboplatin; Magnetic Resonance Spectroscopy; X-Rays

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (chemotherapy, STEMVAC, GM-CSF) (Experimental): See Detailed Description.
  Interventions: Biological: CD105/Yb-1/SOX2/CDH3/MDM2-polyepitope Plasmid DNA Vaccine; Drug: Cisplatin; Procedure: Computed Tomography; Procedure: Computed Tomography Assisted Biopsy; Drug: Docetaxel; Drug: Doxorubicin; Drug: Eribulin; Drug: Paclitaxel; Drug: Pegylated Liposomal Doxorubicin Hydrochloride; Biological: Sargramostim; Procedure: Ultrasound-Guided Biopsy; Procedure: Biospecimen Collection; Drug: Carboplatin; Procedure: Positron Emission Tomography (PET)

INTERVENTIONS:
Biological: CD105/Yb-1/SOX2/CDH3/MDM2-polyepitope Plasmid DNA Vaccine — Given ID
  Other Names: CD105/Yb-1/SOX2/CDH3/MDM2 Plasmid Vaccine; STEMVAC; STEMVAC Th1 Polyepitope Plasmid-based Vaccine
Drug: Cisplatin — Given cisplatin
  Other Names: Abiplatin; Blastolem; Briplatin; CDDP; Cis-diammine-dichloroplatinum; Cis-diamminedichloridoplatinum; Cis-diamminedichloro Platinum (II); Cis-diamminedichloroplatinum; Cis-dichloroammine Platinum (II); Cis-platinous Diamine Dichloride; Cis-platinum; Cis-platinum II; Cis-platinum II Diamine Dichloride; Cismaplat; Cisplatina; Cisplatinum; Cisplatyl; Citoplatino; Citosin; Cysplatyna; DDP; Lederplatin; Metaplatin; Neoplatin; Peyrone's Chloride; Peyrone's Salt; Placis; Plastistil; Platamine; Platiblastin; Platiblastin-S; Platinex; Platinol; Platinol- AQ; Platinol-AQ; Platinol-AQ VHA Plus; Platinoxan; Platinum; Platinum Diamminodichloride; Platiran; Platistin; Platosin
Procedure: Computed Tomography — Undergo CT scans
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; tomography
Procedure: Computed Tomography Assisted Biopsy — Undergo CT-guided biopsy
  Other Names: Computed Tomography Biopsy; Computed Tomography-Guided Needle Biopsy; CT Assisted Biopsy; CT Guided Biopsy
Drug: Docetaxel — Given docetaxel
  Other Names: Docecad; RP 56976; RP-56976; RP56976; Taxotere; Taxotere Injection Concentrate
Drug: Doxorubicin — Given doxorubicin
  Other Names: Adriablastin; Hydroxydaunomycin; Hydroxyl Daunorubicin; Hydroxyldaunorubicin
Drug: Eribulin — Given eribulin
  Other Names: E 7389; E-7389; ER 086526; ER-086526; ER086526
Drug: Paclitaxel — Given paclitaxel
  Other Names: Anzatax; Asotax; Bristaxol; Praxel; Taxol; Taxol Konzentrat
Drug: Pegylated Liposomal Doxorubicin Hydrochloride — Given liposomal doxorubicin
  Other Names: ATI-0918; Caelyx; Dox-SL; Doxil; Doxilen; Doxorubicin HCl Liposomal; Doxorubicin HCl Liposome; Doxorubicin Hydrochloride Liposome; Duomeisu; Evacet; LipoDox; Lipodox 50; Liposomal Adriamycin; Liposomal Doxorubicin Hydrochloride; Liposomal-Encapsulated Doxorubicin; Pegylated Doxorubicin HCl Liposome; Pegylated Liposomal Doxorubicin; S-Liposomal Doxorubicin; Stealth Liposomal Doxorubicin; TLC D-99
Biological: Sargramostim — Given ID
  Other Names: 23-L-Leucinecolony-Stimulating Factor 2; DRG-0012; Leukine; Prokine; rhu GM-CFS; Sagramostim; Sargramostatin
Procedure: Ultrasound-Guided Biopsy — Undergo ultrasound-guided biopsy
  Other Names: Ultrasound Biopsy; Ultrasound Guided Biopsy
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection
Drug: Carboplatin — Given carboplatin
  Other Names: Blastocarb; Carbosin; Carbosol; CBDCA; Displata; Ercar; JM-8; JM8; Nealorin; Novoplatinum; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
Procedure: Positron Emission Tomography (PET) — Undergo PET scan
  Other Names: Medical Imaging; PET scan; PT

SUMMARY:
This phase II trial studies how well a cancer vaccine called STEMVAC works in combination with chemotherapy in treating patients with PD-L1 negative, triple-negative breast cancer that has spread from where it first started (primary site) to other places in the body (metastatic). STEMVAC is designed to target proteins that are expressed on breast cancer stem cells, and it is believed to work by boosting the immune system to recognize and destroy the invader tumor cells that are causing the disease. The allowable combination chemotherapy includes: (1) Paclitaxel is in a class of chemotherapy medications called antimicrotubule agents. It stops tumor cells from growing and dividing and may kill them. (2) Docetaxel is in a class of chemotherapy medications called taxanes. It stops tumor cells from growing and dividing and may kill them. (3) Cisplatin is in a class of chemotherapy medications known as platinum-containing compounds. It works by killing, stopping or slowing the growth of tumor cells. (4) Carboplatin is in a class of chemotherapy medications known as platinum-containing compounds. It works in a way similar to the anticancer drug cisplatin but may be better tolerated than cisplatin. Carboplatin works by killing, stopping or slowing the growth of tumor cells. (5) Doxorubicin is in a class of chemotherapy medications called anthracyclines. Doxorubicin damages the cell's deoxyribonucleic acid (DNA) and may kill tumor cells. It also blocks a certain enzyme needed for cell division and DNA repair. (6) Liposomal doxorubicin is a form of the anticancer drug doxorubicin that is contained inside very tiny, fat-like particles. Liposomal doxorubicin may have fewer side effects and work better than other forms of the drug. (7) Eribulin is in a class of chemotherapy medications called microtubule dynamics inhibitors. It works by stopping the growth and spread of tumor cells. Giving STEMVAC in combination with chemotherapy may be an effective treatment for PD-L1 negative metastatic triple-negative breast cancer.

DETAILED DESCRIPTION:
OUTLINE:

Patients receive one of the following chemotherapy regimens, per the treating physician's discretion, in the absence of disease progression or unacceptable toxicity: 1) Paclitaxel every 21 days; paclitaxel on days 1, 8, and 15 every 28 days; paclitaxel on days 1 and 8 every 21 days; or docetaxel every 21 days; 2) Carboplatin every 21 days; carboplatin every 28 days; carboplatin on days 1 and 8 every 21 days; or cisplatin every 21 days; 3) Doxorubicin every 21 days; or liposomal doxorubicin every 28 days; OR 4) Eribulin on days 1 and 8 every 21 days. Patients receive 3 priming doses of STEMVAC with sargramostim intradermally (ID) every 21-28 days (7-10 days after each chemotherapy administration or during the off week of weekly chemotherapy), 2 booster STEMVAC/sargramostim doses at 4 and 7 months after 3rd priming dose, and then every 6 months in the absence of disease progression or unacceptable toxicity. Patients also undergo computed tomography (CT) or ultrasound-guided biopsy, for research purposes, on study, as well as CT or positron emission tomography (PET) scans and blood sample collection throughout the study. In addition, patients may also undergo CT or ultrasound-guided biopsy, for research purposes, during screening.

After completion of study treatment, patients are followed up at 21 or 28 days and then every 6 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be at least ≥ 18 years of age

  * Note: Because no dosing or adverse event (AE) data are currently available on the use of STEMVAC in patients < 18 years of age, children and adolescents are excluded from this study, but will be eligible for future pediatric trials, if applicable
* Patients with Eastern Cooperative Oncology Group (ECOG) Performance Status Score of ≤ 2
* Histologically confirmed triple-negative breast cancer

  * Tumors with estrogen receptor (ER)-low (≤ 5%) or negative and progesterone receptor (PR)-low (≤ 5%) or negative will be included
  * HER2-negative or HER2-low will be fined by the American Society of Clinical Oncology (ASCO)/College of American Pathologists (CAP) 2023 "Human Epidermal Growth Factor Receptor 2 (HER2) Breast Testing Guideline Update" which reaffirms the 2018 "HER2 Breast Testing Guideline Focused Update"
* Tumor is negative for PD-L1 marker testing per standard of care antibodies/clones in breast cancer at time of eligibility
* Metastatic disease that is measurable based on Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 or PET Response Criteria in Solid Tumors (PERCIST). Target lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions
* Have at least 1 site of disease confirmed by the treating oncologist that could be biopsied during treatment. This site should not be a site that is used to determine measurable disease for efficacy purposes. Lesions that will be biopsied should not be in a previously irradiated area unless progression has been demonstrated in such lesions
* Patients should not have received any prior cancer immunotherapy in the metastatic setting
* Prior Food and Drug Administration (FDA)-approved antibody drug conjugates are allowed
* Patients are appropriate candidates to receive standard of care chemotherapy as per treating oncologist's clinical judgement

  * NOTE: Only chemotherapy partners listed in the protocol are allowed to be administered in metastatic setting concurrently with STEMVAC vaccine
* Patients who have received prior neoadjuvant or adjuvant chemotherapy are allowed
* A minimum of 14 days washout since last systemic therapy or any palliative radiotherapy is required
* Treatment with a bisphosphate or denosumab concurrently with protocol-specific therapy is allowed while on study (it is not exclusionary)
* Patients must be at least 28 days post systemic steroids prior to enrollment, unless this is a steroid administered concurrently with chemotherapy or used as part of prophylaxis to prevent intravenous (IV) contrast reactions
* Must have recovered from major infections and/or surgical procedures; and in the opinion of the investigator, not have any significant active concurrent medical illnesses or condition precluding protocol treatment
* Willing to undergo up to two serial biopsies while on study
* White blood cell (WBC) ≥ 2500/mm^3 (Within 28 days of receiving first study vaccine)
* Lymphocyte count ≥ 500/mm^3 (Within 28 days of receiving first study vaccine)
* Absolute neutrophil count (ANC) ≥ 1000/μL (Within 28 days of receiving first study vaccine)
* Hemoglobin (Hgb) ≥ 9 g/dl (Within 28 days of receiving first study vaccine)
* Platelets ≥ 75,000/μL (Within 28 days of receiving first study vaccine)
* Total bilirubin ≤ 1.5 x institutional upper limit of normal (ULN), except patients with Gilbert's syndrome in whom total bilirubin must be < 3.0 mg/dL (Within 28 days of receiving first study vaccine)
* Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) ≤ 1.5 X institutional ULN (Within 28 days of receiving first study vaccine)
* Creatinine ≤ 1.5 X ULN mg/dL or creatinine clearance > 60 ml/min (Within 28 days of receiving first study vaccine)
* Patients of child-bearing potential must agree to use dual methods of contraception and have a negative urine pregnancy test at screening, and male patients must use an effective barrier method of contraception if sexually active with a person of child-bearing potential. Acceptable methods of contraception are abstinence, condoms with contraceptive foam, oral, implantable or injectable contraceptives, contraceptive patch, intrauterine device, diaphragm with spermicidal gel, or a sexual partner who is surgically sterilized or post-menopausal. Effective methods of contraception must be used throughout the study until the end of treatment on study

Exclusion Criteria:

* Patient has received more than one line of prior therapy in metastatic setting
* Patients with tumors that are PD-L1-positive
* Enrollment in a concurrent interventional clinical trial. Biomarker or tissue collection or any other non-interventional clinical trial enrollment is allowed
* Patients with any of the following cardiac conditions:

  * Symptomatic restrictive cardiomyopathy
  * Dilated cardiomyopathy
  * Unstable angina within 4 months prior to enrollment
  * New York Heart Association functional class III-IV heart failure on active treatment
  * Symptomatic pericardial effusion
* Patients with any autoimmune disease or comorbidities requiring chronic steroids or immunosuppressants
* Known hypersensitivity reaction to the granulocyte-macrophage colony stimulating factor (GM-CSF) adjuvant; any known contra-indication to GM-CSF
* A non-breast malignancy requiring radiation or systemic therapy within last 5 years
* Pregnant and breastfeeding individuals
* Known history of human immunodeficiency virus (HIV) infection, hepatitis B (e.g., hepatitis B virus surface antigen [HBsAg] reactive), or hepatitis C (e.g., hepatitis C virus [HCV] ribonucleic acid [RNA] [qualitative] is detected)
* Major surgery within the 4 weeks prior to initiation of study vaccine
* Must be 14 days between a non-study and non-live vaccine and any STEMVAC vaccination

  * Note: The minimum of 14 days does not apply to the tetanus and diphtheria (Td) vaccine
* Any condition that may interfere with the patient's participation in the study per treating physician

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2027-04-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | From the start of treatment to the worsening of cancer or death whichever occurs first, assessed up to 3 years after completion of study treatment
  Assessed by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1/Positron Emission Tomography (PET) Response Criteria in Solid Tumors (PERCIST).
  Kaplan-Meier method will be used to estimate PFS and the rates at specified time point (e.g., 6 or 12 months) will be calculated and the 95% confidence intervals will be provided.

SECONDARY OUTCOMES:
Overall survival (OS) | Up to 3 years after completion of study treatment
  Kaplan-Meier method will be used to estimate OS and the rates at specified time point (e.g., 6 or 12 months) will be calculated and the 95% confidence intervals will be provided.
Incidence of adverse events | Up to 21 or 28 days after completion of study treatment
  Will be determined by chemical and clinical parameters evaluated at various time points. Toxicity grading will be evaluated according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events version 6.0 and monitoring of adverse events will be done per Food and Drug Administration and NCI guidelines. Descriptive statistics will be provided on the key demographic and clinical variables, such as mean, standard deviation, and range for continuous variables, and percent and number for categorical variables, such as toxicity grades.
Immunogenicity of CD105/Yb-1/SOX2/CDH3/MDM2-polyepitope plasmid deoxyribonucleic acid vaccine (STEMVAC) | Baseline up to 7 months after STEMVAC priming dose #3
  Defined as the sum of the interferon gamma enzyme-linked immunosorbent spot of all STEMVAC antigens on blood samples collected pre-vaccine as compared to 1-month post dose #3 of the STEMVAC vaccine and again after 2 booster doses of STEMVAC vaccine. Both incidence and magnitude will be assessed. Will generate boxplots for its measurements at different timepoints (pre-vaccine, 1 month after vaccine 3, and at each booster) and spaghetti plots to show the changes over time. To make the full use of longitudinal data, will use a weighted generalized estimating equation approach to assess the association between the longitudinal measures over time and a covariate of interest.

CONTACTS AND LOCATIONS:
Overall Officials: Mary Disis, MD, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No